CLINICAL TRIAL: NCT04906226
Title: The Effect of Self-Foot Massage on Peripheral Neuropathic Pain, Peripheral Skin Temperature and Patient Comfort in Diabetic Individuals: A Randomized Controlled Trial
Brief Title: Effect of Self-Foot Massage on Diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, KADRİYE SAYIN KASAR, PhD, RN, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-020
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 diabetes; Foot massage; Neuropathic pain; Skin temperature; Comfort
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Neuralgia

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals participating in the study will be divided into intervention and control groups. The individuals in the foot massage group will be given foot massage training by the researcher. Later, people with diabetes will be enabled to continue self-massage at home. To encourage the continuation of the intervention, the researcher will be called once a week by phone and her questions will be answered. At the end of the four weeks, the patient will be interviewed again and data collection forms will be filled.
  Interventions: Behavioral: Self-foot massage
- Control group (No Intervention): There will be no additional application other than routine to the control group, data collection forms will be applied and recorded at the beginning of the study and at the end of four weeks.

INTERVENTIONS:
Behavioral: Self-foot massage — The individuals in the foot massage group will be given foot massage training by the researcher. Later, people with diabetes will be enabled to continue self-massage at home. To encourage the continuation of the intervention, the researcher will be called once a week by phone and her questions will be answered. At the end of the four weeks, the patient will be interviewed again and data collection forms will be filled.
  Arms: Intervention group

SUMMARY:
The aim of this study is to evaluate the effect of self-foot massage on peripheral neuropathic pain, peripheral skin temperature and patient comfort in individuals with diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is the most important metabolic disease that can affect almost every organ system in the body. Although diabetes causes many macrovascular and microvascular complications, one of the rare microvascular complications is peripheral neuropathy. One of the common complementary and integrative applications in the management of diabetic peripheral neuropathy is foot massage. The aim of this study is to evaluate the effect of self-foot massage on peripheral neuropathic pain, peripheral skin temperature and patient comfort in individuals with diabetes. Individuals participating in the study will be divided into intervention and control groups. The individuals in the foot massage group will be given foot massage training by the researcher. Later, people with diabetes will be enabled to continue self-massage at home. To encourage the continuation of the intervention, the researcher will be called once a week by phone and her questions will be answered. There will be no additional application other than routine to the control group, data collection forms will be applied and recorded at the beginning of the study and at the end of four weeks. In the collection of data, "Individual Description Form, Visuel Analog Scale- (VAS), DN4 Pain Questionnaire and General Comfort Questionnaire- Short form" will be used. In addition, peripheral skin temperature will be measured with a skin thermometer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above,
* Having been diagnosed with type 2 diabetes at least 6 months ago,
* HbA1c level> 6.5%,
* Being able to do personal care for personal hygiene management,
* No peripheral circulation problems,
* Do not have any problems such as speech or hearing that prevent communication,
* Physical and cognitive health levels are suitable for answering the data collection form,
* Agreeing to participate in the research,
* It is planned to include patients who can speak and understand Turkish.

Exclusion Criteria:

* Individuals with other health problems that may cause peripheral neuropathy (chemotherapy, neurological, etc.),
* Patients with organ damage (gangrene or foot / finger amputation) due to diabetes mellitus or any other reason, malignancy, tuberculosis, asthma, or any contagious disease,
* Individuals with a history of disease that may cause changes in peripheral skin temperature (Raynaud's disease, etc.)
* Who do not agree to participate in the research,
* Speaking and hearing impairments that interfere with the collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale- (VAS) | 1 months
  The Visual Analogue Scale (VAS), which is used for the assessment of pain, is used to convert some values that cannot be measured numerically into numerical ones.
DN4 Pain Questionnaire | 1 months
  The DN4 pain questionnaire is a questionnaire that includes symptoms and signs associated with neuropathic pain.
General Comfort Questionnaire- Short form | 1 months
  It is used to determine the comfort level of patients.
Peripheral skin temperature will be measured with a skin thermometer | 1 months
  The skin temperature in the middle of the plantar surfaces of both feet is measured using the handheld digital skin thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye SAYIN KASAR, PhD, RN, Principal Investigator — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No